CLINICAL TRIAL: NCT06274970
Title: PaThERAS Study- Application of Enhanced Recovery After Surgery Protocols in Thyroid and Parathyroid Surgery
Brief Title: PaThERAS: ERAS Protocols in Thyroid & Parathyroid Surgery
Acronym: PaThERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Gaurav Agarwal, Professor and Head of Department Endocrine and Breast Surgery, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-143-Mch-EXP-50
Record Dates: First submitted 2024-01-16; First posted 2024-02-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Diseases; Parathyroid Diseases; ERAS
Keywords: ERAS Protocols; Enhanced Recovery After Surgery Protocols; Thyroid Surgery; Parathyroid Surgery; PaThERAS
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERAS Group (Experimental): Those patients who follow ERAS protocols preoperatively, intraoperatively and post operatively
  Interventions: Other: Enhanced recovery protocols
- Conventional Group (Active Comparator): Those patients who conventional protocols preoperatively, intraoperatively and post operatively
  Interventions: Other: Conventional Protocols

INTERVENTIONS:
Other: Enhanced recovery protocols — Aforementioned in the detailed description
  Arms: ERAS Group
Other: Conventional Protocols — Conventional protocols for non-ERASP group Eg: No preoperative vitamin D and calcium supplementation etc.
  Arms: Conventional Group

SUMMARY:
Enhanced recovery after surgery (ERASP) are evidence-based perioperative protocols devised to expedite postoperative recovery and discharge, decrease surgical stress and costs. However, there is limited data on their use and effectiveness in thyroid and parathyroid surgery. Aim of PaThERAS study is to investigate the clinical benefits and cost-effectiveness of enhanced recovery protocols for the perioperative management in patients undergoing total thyroidectomy for large goiters/ cancers and parathyroidectomy for symptomatic hyperparathyroidism in non-day-care setting.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES

AIM: To evaluate if Enhanced recovery after surgery protocols; improves peri-operative outcomes in patients undergoing thyroid and parathyroid surgery

OBJECTIVES:

Primary Objective: To compare the rate of hypocalcemia in patients undergoing thyroid and parathyroid surgery implementing Enhanced recovery after surgery protocols vs Conventional peri operative protocols Secondary Objective: To compare the following outcome measures in in patients undergoing thyroid and parathyroid surgery

* length of hospital stay- defined as length of hospital stay from the date of surgery to the date of discharge
* hospital costs
* readmission rate
* postoperative complication rates

MATERIALS AND METHODS

1. Study area: This study will be conducted in the Department of Endocrine and Breast Surgery of Sanjay Gandhi Post Graduate Institute, Lucknow, India
2. Study design: The present study will be a prospective study (Amendment to previous protocol was approved by Institutional Ethics Committee)

   * Study group: Prospective cohort
   * Control group: Prospective cohort
3. Study Population:

   Study group (Group 1)
   * Consecutive patients undergoing thyroid and parathyroid surgery in the Dept of Endocrine and Breast Surgery, SGPGI, consenting to participate in the study Control group (Group 2)
   * Screening and review of clinical data from the HIS & patient files
   * All age and sex matched patients who underwent similar procedures from Jan 2021-Sept 2024
4. Inclusion Criteria: Patients diagnosed to have ASA Grade 1 and Grade 2 patients with thyroid and/or parathyroid (1° and 2° hyperparathyroidism) disease undergoing the following procedures via open or endoscopic approach

   • Total thyroidectomy/Focused parathyroidectomy/BNE with excision of enlarged glands +/- any additional procedure (Eg: Central compartment neck dissection, Lateral neck dissection, Cervical thymectomy etc)
5. Exclusion Criteria: Patients undergoing thyroid and/or parathyroid surgery who

   * Undergo hemithyroidectomy
   * Refuse to consent to participate in the study in the cohort group
   * ASA Grade 3 and Grade 4* *Comorbidities of severe nature which may independently impact perioperative hospital stay, complications and outcomes in the study and control group
6. Sample Size

   * Primary objective -To compare the LOS in patients implementing enhanced recovery protocols versus conventional perioperative practices in thyroid and parathyroid surgery
   * Considering the hospital stay to be 5 days in the control group and 3.5 days in the study group (expecting at least 30% reduction in hospital stay); the standard deviation (SD) being 2.5 days and 1.75 days respectively (assuming 50% SD of mean) at minimum one-sided Confidence interval and 95% Power of study- the study requires 44 patients each in the control group and the intervention group
   * Sample size was calculated using software PASS 16
7. Study period: Jan 2023- to Sept 2024

   METHODOLOGY This study is being undertaken after approval by the Institutional Ethics committee. This is a prospective study on all patients undergoing thyroid and/or parathyroid surgery who meet the inclusion criteria admitted in the Department of Endocrine Surgery ward, SGPGI, Lucknow. Each patient in the study will be identified using stickers on their file and OPD booklet/card as SGPGI Endocrine Surgery ERASP patients

   Selection of subjects

   Outcome measures: Those patients diagnosed as having either benign or malignant thyroid and/or parathyroid disease will be enrolled after taking an informed consent. In patients implementing enhanced recovery protocols versus conventional perioperative practices the following outcomes will be compared:
   * The length hospital of stay- Date of surgery to date of discharge = no. of days from date of surgery to date of discharge
   * Hospital costs- Absolute Billing Amount including hospital stay rental, investigations, medications & consumables, and surgical fees (minus) Preoperative stay room rent charges
   * Postoperative complication rates:

     * Hypocalcemia- defined as corrected S. Calcium levels <8.0mg/dl on Post operative day (POD) 1, POD2, POD7-10
     * Surgical site infection- Incisional infection within 30 days after surgery and at least one of the following-

       * Purulent drainage, with/without lab confirmation from the superficial incision
       * Organisms isolated from aseptically obtained culture fluid or tissue from the superficial incision
       * At least one of the following signs or symptoms of infection pain or tenderness, localised swelling, erythema, heat and superficial incision is deliberately opened by the surgeon in a culture negative wound
     * Seroma- Accumulation of clear fluid in a tissue or body cavity (will be assessed after drain removal)
     * Hematoma- Accumulation of blood in a tissue or body cavity (will be assessed daily until discharge)
     * Pain - Measured on Numeric Pain Rating Scale daily until discharge
   * Readmission rate- Number of readmissions after discharge The steps followed in the Enhanced recovery protocol were based on adaptations from recommendations by the ERAS society guidelines on head and neck surgery with free flap reconstruction and literature including meta-analyses and systematic reviews as well as randomized controlled trials wherever possible. In the absence of high level data, case series and nonrandomized studies, ATA statements in thyroid and parathyroid surgeries were considered. These recommendations were adapted and modified to make an Institutional Enhanced recovery protocol to cater to the Indian/South Asian demography. Critical team members include the OPD team, operating surgeon, OT team, anesthesiologist, and ward team and ward nursing staff.

   Enhanced recovery Protocol Recommendation

   Preoperative Considerations Preadmission education- All patients undergoing thyroid and parathyroid surgery will be counselled by a study team member and handed over the study patient information sheet for all information on what to expect before and after surgery

   Perioperative nutritional care- All patients undergoing thyroid and parathyroid surgery should undergo preoperative nutritional assessment Grading of Nutritional Status of the patient (BMI) in kg/m2

   Peri operative Calcium and Vitamin D supplementation-The role for perioperative vitamin D supplementation in preventing symptoms has been studied at length and shown to be beneficial. All Patients with preoperative Vitamin D levels <45nmol/L will be administered loading dose of Cholecalciferol 60k IU/gm for 5 days followed by once a month. Post operatively patients will be prophylactically started on 2g of oral Calcium carbonate tablets, Calcitriol supplementation +/- Parenteral Calcium supplementation only if symptomatic for hypocalcemia or pre-tetany (Trousseau's sign /Chovstek's sign positive)

   Preoperative fasting should be minimized Prior to anaesthesia -Clear fluids should be permitted for up to 2 hours and solids for up to 6 hours. Carbohydrate loading clear drink 180ml (180ml= 1glass) administered to the patient at 6:00 AM in the morning of surgery along with medicines as prescribed by the Anaesthesiologist Oral diet is the first choice for all patients tolerating it Nutrition interventions should be developed in consultation with the multidisciplinary team and individualized according to nutritional status and surgical procedure.

   Antibiotic prophylaxis- Perioperative antibiotics are not indicated for short clean procedures.

   Single dose prophylactic broad spectrum antibiotic is administer intravenously at the time of anesthesia induction/ within 1 hour of incision. Dose is repeated if operative time exceeds 4 hours.

   Choice of antibiotic- 6-monthly rotational/ alternating practice, as per Hospital infection control committee policy is used. Inj. Amoxycillin 1g + Potassium Clavulanate 200mg (1.2gm) OR Inj. Cefuroxime 1.5gms is administered. In patients with hypersensitivity to either of these, an appropriate substitute e.g. Fluroquinolones like Inj. Ciprofloxacin 400mg is administered.

   Postoperative nausea and vomiting prophylaxis- Patients undergoing thyroid and parathyroid surgery should receive preoperative medications to prevent postoperative nausea and/or vomiting.

   Tab Pantoprazole 40mg HS and morning of surgery - All ASA Grade 1 and 2 patients are to take their premedication with 1 glass (180 ml) of Carbohydrate loading clear drink at 6:00 AM in the morning of surgery

   Pre anaesthetic medications- Patients should receive short acting anxiolytics, given intravenously and titrated to required effect. Longer acting anxiolytics and opioids should be avoided.

   Tab. Alprazolam 0.25mg will be given HS and on the morning of surgery

   Skin preparation Chlorhexidine bath on the night prior to and morning of surgery On table part preparation with Chlorhexidine 4% solution/ Povidone-Iodine 10% solution. Prep must be allowed to air dry (minimum 3 minutes) before draping and incision

   Operative Considerations Preventing hypothermia Normothermia should be maintained intraoperatively. Temperature monitoring is necessary to ensure normothermia is maintained.

   Patient adequately covered after placement of ECG leads (use warmer) Warmer used Warm Fluids used at ALL time Head adequately covered (especially in children) Hot line used wherever appropriate Always aim for >36 degrees C temperature

   Perioperative fluid management- Fluids should be managed in a goal-directed manner, avoiding over and under hydration. No fluids should be administered in preop room. Discontinue IV fluids once patient can tolerate orally >500ml or 4-6 hours post extubation

   Intra operative Nerve monitoring (IONM)- Laryngeal nerve monitoring will be used as per operating surgeon's discretion Long-acting neuro muscular blockade should be avoided if IONM is being used

   Dressings and drain use- Pressure dressings do not prevent postoperative hematoma, and may obscure visualization of a hematoma. Several randomized prospective studies have shown that the use of a drain after uncomplicated total thyroidectomy, lobectomy, and subtotal thyroidectomy likewise does not reduce the rate of postoperative bleeding Patient will be discharged with drain once there are no signs of bleeding in the drain or after drain removal if drain out put <20ml/day

   Post operative Considerations Pain management Opioid-sparing, multimodal analgesia, utilizing NSAIDs and paracetamol, are preferred Pain will be assessed using Numeric Pain Rating Scale Inj Paracetamol 1gm iv TDS will be administered until the patient is able to tolerate orally Once the patient is orally allowed -Tab Paracetamol 650mg po TDS will be administered if pain 0-3-mild on Numeric Pain Rating Scale. If Pain on Numeric Pain Rating Scale >/= 4 SOS NSAIDS will be added

   Postoperative mobilization- Early mobilization, within the first 24 hours of surgery is recommended

   Urinary catheterization- Urinary catheters are ordinarily inserted only if anticipated duration of surgery is >4 hours. Urinary catheters should be removed as soon as the patient is able to void, ideally less than24 hours after completion of surgery

   Postoperative pulmonary physical therapy-Pulmonary physical therapy should be initiated as early as possible after surgery to avoid pulmonary complications.

   Head of bed elevation to 30 degrees Steam Inhalation 5 mins thrice daily Incentive spirometry 15 repetitions every 2 hours when the patient is awake Chest Physiotherapy - Attendant/nurse/doctor using cupped hands, Thumping/percussion of posterior lung fields for 5 mins thrice daily

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have ASA Grade 1 and Grade 2 patients with thyroid and/or parathyroid (1° and 2° hyperparathyroidism) disease undergoing the following procedures via open or endoscopic approach • Total thyroidectomy/Focused parathyroidectomy/BNE with excision of enlarged glands +/- any additional procedure (Eg: Central compartment neck dissection, Lateral neck dissection, Cervical thymectomy etc)

Exclusion Criteria:

* Patients undergoing thyroid and/or parathyroid surgery who

  * Undergo hemithyroidectomy
  * Refuse to consent to participate in the study in the cohort group
  * ASA Grade 3 and Grade 4* *Comorbidities of severe nature which may independently impact perioperative hospital stay, complications and outcomes in the study and control group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
To compare the rate of hypocalcemia in patients undergoing thyroid and parathyroid surgery implementing Enhanced recovery after surgery protocols vs Conventional peri operative protocols | Post operative day 1, 2 & 7
  S. Calcium levels will be measured. Levels >8mg/dl were considered normal

SECONDARY OUTCOMES:
To compare length of hospital stay in patients undergoing thyroid and parathyroid surgery in days | from date of surgery till Post operative Day 7
  length of hospital stay defined as length of hospital stay in days from the date of surgery to the date of discharge
To compare hospital costs in patients undergoing thyroid and parathyroid surgery implementing Enhanced recovery after surgery protocols vs Conventional peri operative protocols | from date of surgery till Post operative Day 7
  In hospital costs will be compared from date of surgery till date of discharge
To compare postoperative complication rates in patients undergoing thyroid and parathyroid surgery implementing Enhanced recovery after surgery protocols vs Conventional peri operative protocols | from date of surgery till 6 months post surgery
  Occurrence of Hematoma, seroma, Surgical site infection,pain
To compare readmission rate | from date of surgery till 6 months post surgery
  Readmissions for any complications related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Agarwal, MS, Principal Investigator — gauravbsi@gmail.com
Locations (1):
- Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Background] Chorath K, Luu N, Go BC, Moreira A, Rajasekaran K. ERAS Protocols for Thyroid and Parathyroid Surgery: A Systematic Review and Meta-analysis. Otolaryngol Head Neck Surg. 2022 Mar;166(3):425-433. doi: 10.1177/01945998211019671. Epub 2021 Jun 15. PMID 34126805
- [Background] Smith TW Jr, Wang X, Singer MA, Godellas CV, Vaince FT. Enhanced recovery after surgery: A clinical review of implementation across multiple surgical subspecialties. Am J Surg. 2020 Mar;219(3):530-534. doi: 10.1016/j.amjsurg.2019.11.009. Epub 2019 Nov 16. PMID 31761300
- [Background] Dort JC, Farwell DG, Findlay M, Huber GF, Kerr P, Shea-Budgell MA, Simon C, Uppington J, Zygun D, Ljungqvist O, Harris J. Optimal Perioperative Care in Major Head and Neck Cancer Surgery With Free Flap Reconstruction: A Consensus Review and Recommendations From the Enhanced Recovery After Surgery Society. JAMA Otolaryngol Head Neck Surg. 2017 Mar 1;143(3):292-303. doi: 10.1001/jamaoto.2016.2981. PMID 27737447
- [Background] Terris DJ, Snyder S, Carneiro-Pla D, Inabnet WB 3rd, Kandil E, Orloff L, Shindo M, Tufano RP, Tuttle RM, Urken M, Yeh MW; American Thyroid Association Surgical Affairs Committee Writing Task Force. American Thyroid Association statement on outpatient thyroidectomy. Thyroid. 2013 Oct;23(10):1193-202. doi: 10.1089/thy.2013.0049. Epub 2013 Sep 14. PMID 23742254
- [Background] Xing T, Hu Y, Wang B, Zhu J. Role of oral calcium supplementation alone or with vitamin D in preventing post-thyroidectomy hypocalcaemia: A meta-analysis. Medicine (Baltimore). 2019 Feb;98(8):e14455. doi: 10.1097/MD.0000000000014455. PMID 30813146
- [Background] Khatiwada AS, Harris AS. Use of pre-operative calcium and vitamin D supplementation to prevent post-operative hypocalcaemia in patients undergoing thyroidectomy: a systematic review. J Laryngol Otol. 2021 Jul;135(7):568-573. doi: 10.1017/S0022215121001523. Epub 2021 Jun 14. PMID 34120662